CLINICAL TRIAL: NCT01965678
Title: Epidemiological Study of Quality of Life in Osteopathy
Acronym: ESoQoLiO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ESoQoLiO-1
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Muscle Skeletal Disorders
Keywords: Osteopathic manipulative treatment; muscle-skeletal disorder; quality of life
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OMT (Experimental)
  Interventions: Other: Osteopathic Manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment

SUMMARY:
Aim of this study is to evaluate the effectiveness of osteopathy in changing quality of life in a large sample of naive patients undergoing osteopathic manipulative treatment.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* affected by muscle-skeletal disorder

Exclusion Criteria:

* younger than 18 years old
* OMT undertaken during the last 12 months
* Any manual therapy received during the last 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in General Health score | baseline and 1 month

SECONDARY OUTCOMES:
change from baseline in Physical Component score | baseline and 1 month
change from baseline in Mental Component score | baseline and 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Accademia Italiana Osteopatia Tradizionale, Pescara, Italy

REFERENCES:
- [Derived] Cerritelli F, Verzella M, Barlafante G. Quality of life in patients referring to private osteopathic clinical practice: a prospective observational study. Complement Ther Med. 2014 Aug;22(4):625-31. doi: 10.1016/j.ctim.2014.05.007. Epub 2014 May 24. PMID 25146065